CLINICAL TRIAL: NCT02224092
Title: Effects of Multivitamin, Multimineral and Phytonutrient Supplementation on Selected Nutrients Blood Level and Heart Health Risk Factors in Russian Population
Brief Title: Effects of Supplementation in Healthy Russian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Collaborators: Russian Institute of Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Amway-2010-RU1
Record Dates: First submitted 2013-12-19; First posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Heart Health Markers; General Nutritional Status
Keywords: heart health; general well-being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Active is a multivitamin multimineral with phytonutrient product.
  Interventions: Dietary Supplement: multivitamin multimineral with phytonutrient supplementation
- Placebo (Placebo Comparator): Placebo is a sugar pill.
  Interventions: Dietary Supplement: multivitamin multimineral with phytonutrient supplementation

INTERVENTIONS:
Dietary Supplement: multivitamin multimineral with phytonutrient supplementation — The multivitamin multimineral with phytonutrient product consists of four tablets per dose, two "Vitamin" tablets, a "Mineral" tablet, and a "Phytonutrient" tablet. The placebo for this trial will be formulated to match the shape and color of all multivitamin multimineral with phytonutrient product tablets, e.g., a Vitamin Placebo, a Mineral Placebo and a Phytonutrient Placebo.
  Other Names: Active is Nutrilite Double X

SUMMARY:
The objectives of this exploratory study are to (1) evaluate the effect of the multivitamin multimineral with phytonutrient product vs. placebo on heart health risk factors following twice-daily consumption for eight weeks; (2) To test the safety and tolerability of the multivitamin multimineral with phytonutrient product vs. placebo following twice-daily consumption for eight weeks.

DETAILED DESCRIPTION:
More and more evidence shows the benefit of fruit and vegetable intake on the maintenance of good health throughout the lift span. Unfortunately, many people in developed and developing societies do not eat a diet with the variety and quantity of fruits and vegetables. Because of this, prevalence of chronic disease increases rapidly in worldwide as well as the burden on the health care system. Therefore, promoting healthy lifestyle and dietary behavior becomes a critical approach in preventing chronic disease development. According to results from the Moscow Behavioural Risk Factor Survey performed from 2000-2001 found that mean fruit and vegetable intake in men and women in Moscow was 190 grams per day, much lower than the World Health Organization's recommended 400 grams per day. This lower than recommended intake would correlate to a lower intake of phytonutrients and antioxidants and may be associated with higher risks for chronic diseases such as cardiovascular disease (CVD) and cancer. In this study, we are particularly interested in understanding whether a multivitamin multimineral with phytonutrient product can improve nutritional status and reduce heart health risk factors in Russian population with low fruit and vegetable intake. This study is conducted in Russia Institute of Nutrition (ION) clinic, which has 200 beds and outpatients department.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy men and women aged from 40 to 70 years of age preferable smokers and who regularly consumes alcohol, and consuming fewer than 12 items found on the Recommended Foods Checklist (see below) per week.
* Individual should be judged to be in good general health on the basis of an interview and abbreviated physical exam.
* Individual understands the procedures and agrees to participate in the study.
* Individual is able and willing to provide written informed consent and confidentiality agreement.

Exclusion Criteria:

* Use of dietary supplements within one week of Day 1. Supplements include any vitamins, minerals, and herbal products, including herbal drinks.
* Presence of cardiovascular disease, hypercholesterolemia, cancer, diabetes mellitus, or any other chronic health condition identified from the findings of the interview.
* Currently treated for uncontrolled hypertension or blood pressure greater > 140 mm Hg systolic or > 90 mm Hg diastolic during seated, resting measurement on two consecutive occasions during visit 1.
* Therapeutic uses of coumadin, aspirin, or other medications that influence hemostasis within four weeks of Day 1.
* Participation in another clinical trial within 30 days of enrollment into the study.
* History or current abuse of drugs or alcohol, or intake > 4 alcoholic beverages per day.
* Known hypersensitivity to study product or any ingredient in study product.
* A change in hormone therapy, including oral contraceptives, within 4 weeks prior to screening, or unwilling to maintain current hormone therapy/oral contraceptive use throughout the course of the study.
* Pregnant or lactating women, or women of child-bearing potential unwilling to use a medically approved form of birth control.
* Any condition that the Principal Investigator believes may put the subject at undue risk.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change of heart risk factors by measuring homocysteine, C reactive protein (CRP), oxidized low-density lipoprotein (Ox-LDL) and lipid profile at baseline and Day 56 | Baseline, Day 56
Change of nutrient status by measuring b-carotene, a- and r-tocopherol, vitamin C, folic acid, B6, B12, zinc, selenium, polyphenols at baseline, Day 28 and Day 56 | Baseline, Day 28 and Day 56

SECONDARY OUTCOMES:
Change of potential heart health risk factors by measuring gamma-glutamyl transferase (GGT) and uric acid | Baseline and Day 56

OTHER OUTCOMES:
Change of anthropomorphic evaluation markers by measuring height, weight, body mass index (BMI, kg/m2), and waist-to-hip ratio at baseline and Day 56 | Baseline and Day 56
Evaluation of general health status, lifestyle and dietary behavior | Baseline
  dietary questionnaire was used.

CONTACTS AND LOCATIONS:
Overall Officials: Vasily A Isakov, M.D., Ph.D., Principal Investigator — Russian Institute of Nutrition
Locations (1):
- Russian Institute of Nutrition, Moscow, Russia